CLINICAL TRIAL: NCT05029284
Title: teleABLE: Adapting a Behavioral Activation-Based Intervention to Reduce Post-Stroke Sedentary Behavior Using Telehealth (Formative Phase)
Brief Title: Behavioral Activation for Post-Stroke Sedentary Behavior Using Telehealth
Acronym: teleABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0059; K23HL159240 (NIH)
Record Dates: First submitted 2021-07-30; First posted 2021-08-31 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Stroke, Ischemic; Stroke Hemorrhagic
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- teleABLE (Experimental): Participants will complete 12 teleABLE sessions via videoconferencing, guided by an intervention therapist and participant workbook.
  Interventions: Behavioral: teleABLE

INTERVENTIONS:
Behavioral: teleABLE — Participants will be guided to self-monitor their daily activities, schedule personally meaningful non-sedentary activities, collaboratively problem solve to overcome barriers to the activity, and self-assess their progress. Participants may be asked to self-monitor their activity levels and complete planned activities between sessions.

SUMMARY:
Adults with stroke-related disability spend more time sedentary than adults without stroke-related disability, which places them at risk for poor cardiovascular health outcomes. Few interventions are designed to reduce post-stroke sedentary time.

The purpose of this research is to test whether the teleABLE (Activating Behavior for Lasting Engagement) Intervention is feasible and acceptable to adults within the first 12 months post-stroke. The hypothesis is that teleABLE can be feasibly delivered using videoconferencing within the first 12 months post-stroke. 10 participants will complete assessments and activity monitoring (activPAL micro3) at 0 (baseline) and 8 (post-intervention)-weeks. Participants will complete 12 sessions of the teleABLE intervention.

Findings from this study will be used to guide the intervention protocol in the planned next phase of this research.

ELIGIBILITY:
Inclusion Criteria:

* Stroke diagnosis ≤12 months prior to study enrollment
* ≥6 hours of sedentary behavior on a typical weekday (assessed by Sedentary Behavior Questionnaire)
* Ambulatory with or without assistive device (assessed by Functional Independence Measure, mobility score ≥5)
* Able to access an electronic device (smartphone, tablet, or computer) that is compatible with a videoconferencing application
* Able to identify a support person with whom the participant has face-to-face interaction at least one time per week
* Able and willing to participate fully in the study and provide informed consent

Exclusion Criteria:

* Currently receiving care in an inpatient rehabilitation, transitional care unit, or skilled nursing facility
* Severe cognitive or communication impairments (inability to respond accurately to complete study telephone screening or complete informed consent)
* Comorbid neurodegenerative disorder (e.g. Parkinson's disease, multiple sclerosis, amyotrophic lateral sclerosis, myasthenia gravis, dementia, Alzheimer's disease, Huntington's disease, glioblastoma)
* Comorbid cancer, currently undergoing chemotherapy or radiation treatment
* Comorbid major depressive disorder (assessed by Patient Health Questionnaire-2, score ≥2)
* Received inpatient treatment or hospitalized for psychiatric condition and/or alcohol or substance abuse within the past 12 months
* Diagnosis of a terminal illness and/or in hospice care
* History of skin sensitivity that precludes the use of medical tape necessary for adherence to activity monitor measure
* Inability to speak, read, or understand English
* Concurrent participation in another rehabilitation intervention research study
* Investigator discretion for safety or adherence reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Kringle, PhD, OTR/L, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | teleABLE
Started | 11
Completed | 10
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | teleABLE
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 53 [40 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: The count of treatment-related serious (e.g. injurious) and non-serious (e.g. fall without injury) adverse events that occur during intervention delivery will be reported.
Time Frame: week 2 through week 7
Measure: Number; unit: adverse events
Arm/Group | teleABLE
Number analyzed (Participants) | 11
adverse events
  Non-serious (e.g., muscle soreness, skin irritation) | 2
  Serious (e.g., injurious fall) | 0

2. Primary Outcome: Participant Satisfaction
Description: Assessed by the Client Satisfaction Questionnaire-8. This is an 8-item questionnaire with each item ranked on an 1 to 4 Likert-type scale. We will compute the mean score across all items. The possible range is 1 to 4, with high scores indicating high satisfaction.
Time Frame: week 8
Measure: Mean (Standard Deviation); unit: score on a scale of 1 to 4
Arm/Group | teleABLE
Number analyzed (Participants) | 10
score on a scale of 1 to 4 | 3.7 (0.3)

3. Secondary Outcome: Change in Participation Restrictions
Description: Assessed by the Activity Card Sort 3. This is a 100-item tool during which participants indicate whether they did the activity prior to their stroke, continue to do the activity since their stroke, or have given up the activity since their stroke. Change in the proportion of activities retained will be reported.
Time Frame: week 0 to week 8
Measure: Median (Inter-Quartile Range); unit: change in % retained activities
Arm/Group | teleABLE
Number analyzed (Participants) | 10
change in % retained activities | 9.5 [-1.5 to 20.5]

4. Secondary Outcome: Change in Health-Related Quality of Life
Description: Assessed by the EuroQol-5 Dimension-5 Level. This is a 5-item self-report questionnaire with each item scored on a 1 to 5 scale. Scores are converted to Index Scores following published procedures (possible range -1 to 1), with high scores indicating high quality of life.
Time Frame: week 0 to week 8
Measure: Median (Inter-Quartile Range); unit: change score on a scale of -1 to 1
Arm/Group | teleABLE
Number analyzed (Participants) | 10
change score on a scale of -1 to 1 | 0.06 [-.01 to 0.11]

5. Secondary Outcome: Change in Sedentary Minutes
Description: Assessed using the activPAL micro3 monitor following a 7-day wear protocol. The mean daily minutes of sitting time accumulated in bouts of 30 minutes or more will be computed for each time point. Change in mean daily minutes of sitting time accumulated in bouts of 30 minutes or more will be reported.
Time Frame: week 0 to week 8
Population: n=1 participant lost to follow-up n=3 participants with <6 valid activPAL days at 1 or more timepoints
Measure: Median (Inter-Quartile Range); unit: change in sedentary minutes
Arm/Group | teleABLE
Number analyzed (Participants) | 7
change in sedentary minutes | 32.2 [-14.3 to 49.8]

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Adverse events were queried using a questionnaire at the Week 8 assessment timepoint. If the treating occupational therapist became aware of an adverse event during an intervention session, it was reported at the time it was discovered.
Arm/Group | teleABLE
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | teleABLE (N=10)
Muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT05029284/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT05029284/ICF_001.pdf